CLINICAL TRIAL: NCT03584815
Title: Is Physiotherapy or Fasciotomy the Best Treatment Option for Chronic Exertional Compartment Syndrome in the Anterior Compartment of the Lower Leg? A Randomized Controlled Trial.
Brief Title: Physiotherapy or Fasciotomy as Treatment for Chronic Exertional Compartment Syndrome in the Lower Leg?
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Bispebjerg Hospital (Other)
Responsible Party: Principal Investigator, Simon Doessing, M.D., PhD, Chief Surgeon. M.D. PhD, Bispebjerg Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: H-18001263
Record Dates: First submitted 2018-06-30; First posted 2018-07-12 (Actual); Last update posted 2023-12-18 (Actual); Status verified 2023-12

CONDITIONS: Compartment Syndrome Nontraumatic Lower Leg
MeSH Terms: interventions — Surgical Procedures, Operative; Fasciotomy; Physical Therapy Modalities

STUDY DESIGN:
Intervention Model Description: Randomized controlled trial
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Surgery/fasciotomy (Active Comparator): Fasciotomy of the anterior and lateral compartments in the lower legs:
  Two linear longitudinal skin incisions, each approximately 4 cm, are made allowing for excision of the fascia in full length. Sharp dissection to the level of the subcutaneous tissues down to the layer of the overlying fascia is performed, and using a finger or blunt instrument, the subcutaneous tissue is swept away from the fascia, so that an unobstructed cut of the fascia can be performed. The fascia overlying the anterior and lateral compartment is meticulously dissected under direct visualization, the fascia is released approximately as far proximal and distal as the muscle belly is. The perimysium is spared.
  Interventions: Procedure: Surgery/Fasciotomy
- Physiotherapy (Active Comparator): 1. Change the running pattern to decrease load on the affected muscles of the lower leg including the eccentric work performed by the tibialis anterior during the rear-foot strike.
  2. Strengthen the major muscles of all lower leg compartments in order address any muscular imbalance/instability around the ankle joint, and to strengthen the main muscle groups responsible for alignment of the hip and knee.
  Interventions: Other: Physiotherapy

INTERVENTIONS:
Procedure: Surgery/Fasciotomy — Open fasciotomy of the anterior and lateral compartment + standard post-operative physiotherapy for 12 weeks
  Arms: Surgery/fasciotomy
Other: Physiotherapy — Intensive physiotherapy for 12 weeks including a change to forefoot/midfoot strike during running
  Arms: Physiotherapy

SUMMARY:
It is hypothesized that physiotherapy including a change in running landing pattern and surgical fasciotomy are equally good as treatment options for chronic exertional compartment syndrome (CECS) of the anterior compartment of the lower leg.

The endpoints/outcomes are:

Change from week 0 (start of study) to week 12 (completion of intervention) in: patient reported outcome measure (PROM) (Exercise induced leg pain Questionnaire (EILP)).

Secondary outcomes are: Visual Analogue Scale (VAS) score after an "exercise provocation test": Change in intracompartmental pressure (ICP)Change in muscle compartment compliance. Change in Global Rating of Change Score/Scale (GRC). Change in Single Assessment Numeric Evaluation (SANE)

The study is important because:

1. Results from recent studies suggest that physiotherapy represents a valid alternative to surgery for the treatment of CECS. Surgery is currently standard treatment and a change towards physiotherapy as primary treatment could potentially reduce both complication rates and costs.
2. Intracompartmental pressure (ICP) is gold standard for diagnosing CECS. However, the association between ICP and symptoms of CECS, both before and after physiotherapeutic and surgical treatment, muscle compartment compliance and intracompartmental perfusion, has not been thoroughly investigated.

DETAILED DESCRIPTION:
CECS of the lower leg is a condition of pain induced by exercise. CECS accounts for 14-33% of lower leg pain in athletes, evenly divided among males and females. Symptoms are described as a tight, cramp like ache that occurs at a well-defined and reproducible point in the exercise bout and increases if the training persists. Relief of symptoms typically occurs within 30 minutes of ending the activity.

The anterior compartment is most commonly affected, followed by the deep posterior, the lateral and the superficial posterior compartment. Often more than one compartment in the same leg is involved, and the condition is reported bilateral in up to 95% of affected athletes.

The pathophysiology of CECS is not fully understood. It is, however, generally agreed that exercise induces abnormal elevation in ICP, which interferes with tissue perfusion and cause painful ischemia affecting the nerves and impairing muscle function. A noncompliant muscle compartment, which is unresponsive to the expansion of muscle volume that occurs with exercise, offer a possible pathophysiological explanation for CECS. However, this view is challenged by a study reporting no difference in fascial thickness and stiffness between CECS patients and healthy controls. Furthermore, the thickness of the anterior compartment increased more with exercise in CECS patients relative to controls, questioning decreased compliance as the main pathophysiology in CECS. The definition of a pathologically elevated ICP during exercise is important for the diagnosis of CECS and is currently debated. The criteria suggested by Pedowitz is used as standard by most clinicians for the diagnosis of CECS: 1) a pre-exercise pressure of 15 mmHg or greater, and/or 2) a 1-minute post-exercise pressure of 30 mmHg or greater, and/or 3) a 5-minute post-exercise pressure of 20 mmHg or greater. The precision and diagnostic value of these commonly used criteria is debated, due to a reported overlap in ICP readings between patients and healthy controls at certain time points. Interestingly, in a small cohort of asymptomatic rollerskiers ICP was elevated, according to the Pedowitz criteria, in 100% of participants after 20 minutes of exercise. Despite these uncertainties, it is suggested that ICP measured 1-minute after ceasing exercise has the highest diagnostic value, as it most consistently display higher values in patients with CECS symptoms relative to healthy controls. The different types of catheters (slid catheter, side-port, straight-needle) also clearly influence the absolute values of the measurements and the catheter tip can be wrongfully placed outside the compartment by experienced health professionals in up to 21% of cases when positioned without ultrasound guidance.

Non-invasive modalities such as magnetic resonance imaging (MRI), near infrared spectroscopy (NIRS) and ultrasound measurements have been suggested as future adjuncts or alternatives for diagnosing CECS, but their diagnostic value remains to be established.

In summary, it is generally agreed that ICP measurements are important for diagnosing CECS, but several studies question current practice including the mentioned criteria and particularly the use of non-ultrasound guided catheter positioning.

Both conservative and surgical treatment options are suggested in the literature.

Conservative treatment, including physiotherapy, has been attempted with varying success and is generally believed by many to be insufficient for the long-term treatment of CECS. However, inducing muscle hypotrophy via injection of botulinum toxin, was efficient in reducing exercise induced pain in CECS patients, but also resulted in decreased muscle strength, although without measurable functional consequences. Interestingly, changing the gait pattern in order to achieve a forefoot/midfoot strike during running, which potentially decrease pressure in the anterior compartment and eccentric load of the anterior compartment muscles has proven successful for treatment of anterior CECS. These studies suggest a role for non-operative treatment of CECS, but to our knowledge, no randomized controlled studies exist regarding the effect of physiotherapy or other non-surgical interventions.

Surgical fasciotomy, with release of the compartment(s) with elevated intra-compartmental pressure, has been shown by many investigators to be effective using both open, mini-open and endoscopically assisted techniques. There are, however, considerable variations in the reported outcomes of surgery. In a large cohort, 45% had symptom recurrence after surgery and 16% experienced surgical complications including infection, neurological damage, and hematoma. Moreover, the need for revision surgery can be as high as 11%. Other groups report more successful outcome of surgery with patient satisfaction of 60 to 90%, including a retrospective follow-up study, in which operation was successful in 81% of patients and non-operative treatment successful in only 41% of patients.

CECS is a common condition in athletes and although disagreements exist, the diagnosis is typically made based on a history of pain in the calf muscles during exercise that resolves within 30 minutes of ending the activity as well as a positive ICP reading. Typically the patients are offered fasciotomy if the symptoms persist.

No studies have compared the effect of fasciotomy to any non-surgical treatment strategies in a randomized controlled setting. Moreover, correlation between symptom severity, ICP measurements, muscle compartment compliance and perfusion, and effect of treatment is not fully elucidated. Finally, the possible effect of changing the landing pattern in combination with physical therapy has not been attempted in a randomized setting.

It is hypothesized that physiotherapy including a change in running landing pattern and surgical fasciotomy are equally good as treatment options for chronic exertional compartment syndrome (CECS) of the anterior compartment of the lower leg.

The endpoints/outcomes are:

Change from week 0 (start of study) to week 12 (completion of intervention) in: patient reported outcome measure (PROM) (Exercise induced leg pain Questionnaire (EILP)).

Secondary outcomes are: Visual Analogue Scale (VAS) score after an "exercise provocation test": Change in intracompartmental pressure (ICP)Change in muscle compartment compliance. Change in Global Rating of Change Score/Scale (GRC). Change in Single Assessment Numeric Evaluation (SANE)

The study is important because:

1. Results from recent studies suggest that physiotherapy represents a valid alternative to surgery for the treatment of CECS. Surgery is currently standard treatment and a change towards physiotherapy as primary treatment could potentially reduce both complication rates and costs.
2. Intracompartmental pressure (ICP) is gold standard for diagnosing CECS. However, the association between ICP and symptoms of CECS, both before and after physiotherapeutic and surgical treatment, muscle compartment compliance and intracompartmental perfusion, has not been thoroughly investigated.

ELIGIBILITY:
Inclusion criteria:

* Age between 18 and 50 years
* Symptoms for more than 3 months
* Symptoms from both legs. Pain (cramp like, tight, burning or pressure) in the anterior part of the lower leg starting after approximately 10 minutes of exercise
* Pain worsened with prolonged lower extremity exertion
* Majority of pain relieved within 30 minutes of rest.

Exclusion criteria:

* Previous fasciotomy in the lower leg
* History of serious trauma involving the lower leg (fracture, muscle/tendon rupture)
* ASA (America Association of Anaesthesiologists Classification of Physical Health) > 2
* Clinical symptoms consistent with unilateral anterior CECS or lateral and posterior CECS
* Clinical symptoms consistent with lumbar spine radiculopathy, periostit/shin-splint, stress fracture, popliteal artery entrapment syndrome, isolated peroneal nerve entrapment, with isolated muscle fascia herniation.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 72 (Estimated)
Dates: Start 2019-05-05 (Actual); Primary Completion 2024-08 (Estimated); Study Completion 2025-08 (Estimated)

PRIMARY OUTCOMES:
Exercise induced leg pain Questionnaire (EILP) | 1 year
  The primary outcome is 10-item uni-dimensional PROM, the "Exercise induced leg pain Questionnaire" (EILP) (Nauck, Lohrer, Padhiar, & King, 2015). Each item is scored on a five point Likert scale from 4 (no difficulty) to 0 (unable to do) with a total score of 40 points. This PROM is developed specifically to quantify the patients perceived severity of exercise induced lower leg symptoms and has a high validity and reliability. We have translated the original German version of the questionnaire into Danish for the purpose of the present study. The translation is in accordance with international standards (Beaton, Bombardier, Guillemin, & Ferraz, 2000) and have been approved by the authors of the original German version.

SECONDARY OUTCOMES:
Intracompartmental pressure (ICP) testing | 12 weeks
  Following treadmill running until symptoms occur with pain reaching 8 on a visual analogue scale (VAS) the patients are positioned supine with a soft pad under the knee, and the knee in 10 degrees flexion and the ankle relaxed in 30 degree plantar-flexion, confirmed with a goniometer. The catheter is inserted at a 90 degree angle with ultrasound guidance to insure correct positioning. To save time, ultrasound is performed before exercise is begun to get the approximate position of the compartments, and the skin is anesthetised, specifically avoiding anesthetizing deep to the skin, using a 23g needle and 0.5% lidocain. Compartment pressure is measured immediately after exercise, after 1-minute and after 5 minutes . We use the handheld Stryker Intracompartmental Monitor System with an 18g side-ported needle (Stryker) as described by Braver. This equipment has proven both accurate and reliable.
Ultrasonic measurement of anterior compartment thickness (ACT) | 12 weeks
  The thickness of the anterior compartment is determined at rest and 0.5 min., 2.5 min., and 4.5 min after treadmill running (described above). The patients are positioned in the same supine position (see above). As described by Rajasekaran (Rajasekaran et al., 2013), ACT is measured at 20% of the distance from the head of the fibula to the lateral tip of the lateral malleolus. The site of measurement is located and marked on the skin prior to exercise provocation. Using Hitachi Avius ultrasound machine (Hitachi Aloka, Tokyo, Japan) with a linear array transducer and general musculoskeletal settings. The ultrasound probe is positioned at an approximated 90-degree angle to the anterior muscle group and parallel to the interosseous membrane. The thickness of the anterior muscle group is determined by measuring the shortest distance from the border of the interosseous membrane facing the anterior compartment and the interior border of the fascia adjacent to the subcutaneous fat.

CONTACTS AND LOCATIONS:
Overall Officials: Simon Doessing, M.D. PhD, Principal Investigator — Institute of Sports Medicine, Bispebjerg Hospital
Locations (2):
- Denmark (2):
  - Bispebjerg Hospital, Copenhagen, Copehagen
  - Bispebjerg Hospital, Copenhagen

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-05-28): https://cdn.clinicaltrials.gov/large-docs/15/NCT03584815/Prot_SAP_000.pdf